CLINICAL TRIAL: NCT05166577
Title: Open-Label Multicenter Phase 1b/2 Study of Nanatinostat + Valganciclovir in Patients With Advanced Epstein-Barr Virus-Positive Solid Tumors and in Combination With Pembrolizumab in Patients With Recurrent/Metastatic Nasopharyngeal Carcinoma
Brief Title: Nanatinostat Plus Valganciclovir in Advanced EBV+ Solid Tumors and in Combination With Pembrolizumab in EBV+ RM-NPC
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Viracta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VT3996-301
Record Dates: First submitted 2021-12-03; First posted 2021-12-22 (Actual); Results first posted 2025-02-24 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-02

CONDITIONS: Nasopharyngeal Carcinoma; EBV-Related Gastric Carcinoma; EBV-Related Leiomyosarcoma; EBV Related Carcinoma; EBV-Related Sarcoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Valganciclovir; pembrolizumab

STUDY DESIGN:
Intervention Model Description: A traditional 3+3 dose escalation design followed first by a dose optimization cohort and then by dose expansion with 1:1 randomization to receive nanatinostat and valganciclovir with or without pembrolizumab in Phase 2.
  The study was prematurely terminated after the end of Phase 1b and did not proceed to Phase 2.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nanatinostat in combination with valganciclovir (Experimental): Phase 1b: Nanatinostat dose escalation starting at 20 mg orally daily, 4 days per week, and valganciclovir starting at 900 mg orally daily, then Phase 2: Nanatinostat and valganciclovir at the confirmed recommended Phase 2 dose
  Interventions: Drug: Nanatinostat; Drug: Valganciclovir
- Nanatinostat in combination with valganciclovir and pembrolizumab (Experimental): Phase 2: Nanatinostat and valganciclovir at the confirmed recommended Phase 2 doses in combination with pembrolizumab 200 mg intravenous (IV) every 3 weeks
  Interventions: Drug: Nanatinostat; Drug: Valganciclovir; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Nanatinostat — Phase 1b: Nanatinostat dose escalation starting at 20 mg orally daily, 4 days per week, then Phase 2: Nanatinostat at the confirmed recommended Phase 2 dose
  Other Names: VRx-3996
Drug: Valganciclovir — Phase 1b: Valganciclovir starting at 900 mg orally daily, then Phase 2: Valganciclovir at the confirmed recommended Phase 2 dose
  Other Names: Valcyte
Drug: Pembrolizumab — Phase 2: Pembrolizumab (anti-PD-1) dosed at 200 mg intravenous (IV) every 3 weeks
  Other Names: Keytruda
  Arms: Nanatinostat in combination with valganciclovir and pembrolizumab

SUMMARY:
This study will evaluate the safety and efficacy of nanatinostat in combination with valganciclovir in patients with relapsed/refractory EBV-positive solid tumors and in combination with pembrolizumab in patients with recurrent/metastatic nasopharyngeal carcinoma

DETAILED DESCRIPTION:
This is an open-label, multicenter Phase 1b/2 study evaluating nanatinostat in combination with valganciclovir alone and in combination with pembrolizumab. Nanatinostat is a selective class I HDAC inhibitor which induces EBV early lytic phase protein generation, activating (val)ganciclovir to its cytotoxic form.

The Phase 1b dose escalation portion is designed to evaluate safety and to determine the recommended Phase 2 dose (RP2D) in patients with EBV+ RM-NPC followed by a Project Optimus | FDA (https://www.fda.gov/about-fda/oncology-center-excellence/project-optimus) cohort to confirm the RP2D. Up to 60 patients with EBV+ RM-NPC will be randomized 1:1 to receive nanatinostat in combination with valganciclovir at the confirmed RP2D with or without pembrolizumab to evaluate safety, overall response rate, and potential pharmacodynamic markers in the Phase 2 dose expansion part of the study. Additionally, patients with other EBV+ solid tumors will be enrolled to receive nanatinostat in combination with valganciclovir at the RP2D in a Phase 1b cohort.

The study was prematurely terminated after the end of Phase 1b and did not proceed to Phase 2.

ELIGIBILITY:
Key Inclusion Criteria:

* Recurrent or metastatic EBV+ nasopharyngeal carcinoma (RM-NPC) for whom no potentially curative options are available, who have received at least 1 prior line of platinum-based chemotherapy and no more than 3 prior lines of therapy for RM-NPC.
* Phase 1b exploratory proof-of-concept cohort only: Advanced/metastatic EBV+ non-NPC solid tumors with no available curative therapies.
* Measurable disease per RECIST v1.1
* ECOG performance status 0 or 1
* Adequate bone marrow and liver function

Key Exclusion Criteria:

* Anti-tumor treatment with cytotoxic drugs, biologic therapy, immunotherapy, or other investigational drugs within 4 weeks or >5 half-lives, whichever is shorter
* Active CNS disease
* Inability to take oral medication, malabsorption syndrome or any other gastrointestinal condition (nausea, diarrhea, vomiting) that may impact the absorption of nanatinostat and valganciclovir
* Active infection requiring systemic therapy
* Active autoimmune disease that has required systemic therapy with modifying agents, corticosteroids, or immunosuppressive agents
* Positive hepatitis B or hepatitis C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-10-08 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2025-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darrel P Cohen, MD, PhD, Study Director — Viracta Therapeutics
Locations (13):
- United States (3):
  - Stanford Cancer Center, Stanford, California
  - University of Colorado Hospital, Aurora, Colorado
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Blacktown Hospital, Blacktown, Australia
- Princess Margaret Cancer Centre, Toronto, Canada
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - Prince Of Wales Hospital, The Chinese University Of Hong Kong, Shatin
- Malaysia (2):
  - Sarawak General Hospital, Kuching, Sarawak
  - University of Malaya Medical Centre, Kuala Lumpur
- National Cancer Centre Singapore, Singapore, Singapore
- Samsung Medical Center, Seoul, South Korea
- Taiwan (2):
  - Taipei Veterans General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Cohort 1: Nanatinostat 20 mg once daily, Days 1-4/week Valganciclovir 900 mg once daily
- Dose Cohort 2: Nanatinostat 30 mg once daily, Days 1-4/week Valganciclovir 900 mg once daily
- Dose Cohort 3: Nanatinostat 40 mg once daily, Days 1-4/week Valganciclovir 900 mg once daily
- Dose Cohort 4: Nanatinostat 10 mg and 10 mg divided dose, Days 1-4/week Valganciclovir 900 mg twice daily x 21 days then once daily
- Dose Cohort 5: Nanatinostat 20 mg and 10 mg divided dose, Days 1-4/week Valganciclovir 900 mg twice daily x 21 days then once daily
- Dose Cohort 6: Nanatinostat 20 mg and 20 mg divided dose, Days 1-7/week Valganciclovir 450 mg twice daily
- Dose Cohort 7: Nanatinostat 20 mg and 10 mg divided dose, Days 1-7/week Valganciclovir 450 mg twice daily
Period: Overall Study
Arm/Group | Dose Cohort 1 | Dose Cohort 2 | Dose Cohort 3 | Dose Cohort 4 | Dose Cohort 5 | Dose Cohort 6 | Dose Cohort 7
Started | 3 | 4 | 3 | 3 | 4 | 3 | 6
Completed | 3 | 4 | 3 | 3 | 4 | 3 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Cohort 1 | Dose Cohort 2 | Dose Cohort 3 | Dose Cohort 4 | Dose Cohort 5 | Dose Cohort 6 | Dose Cohort 7 | Total
Number analyzed (Participants) | 3 | 4 | 3 | 3 | 4 | 3 | 6 | 26
Age, Continuous [Mean (Full Range); unit: Years] | 43 [19 to 61] | 52 [44 to 59] | 42 [33 to 48] | 54 [33 to 66] | 51 [39 to 63] | 48 [44 to 56] | 55 [41 to 69] | 50 [19 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 0 | 0 | 2 | 2 | 5
  Male | 3 | 4 | 2 | 3 | 4 | 1 | 4 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 3 | 3 | 3 | 3 | 3 | 5 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Black or African American | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 3
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumor Type [Count of Participants; unit: Participants]
  EBV+ Nasopharyngeal Carcinoma | 3 | 4 | 3 | 3 | 4 | 3 | 6 | 26
  Other EBV+ Cancer | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Incidence of Dose-Limiting Toxicities (DLTs)
Description: Percentage of patients experiencing a DLT, defined as an adverse event or clinically significant abnormal laboratory value that is at least possibly related to study drugs and is not primarily related to disease, disease progression, concomitant medication(s), or intercurrent illness
Time Frame: DLT period of 28 days
Population: Phase 1b safety analysis population, defined as all patients with recurrent or metastatic EBV+ nasopharyngeal carcinoma who received at least one dose of study treatment in Phase 1b
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Cohort 1 | Dose Cohort 2 | Dose Cohort 3 | Dose Cohort 4 | Dose Cohort 5 | Dose Cohort 6 | Dose Cohort 7
Number analyzed (Participants) | 3 | 4 | 3 | 3 | 4 | 3 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 2 | 0

2. Primary Outcome: Phase 2: Overall Response Rate (ORR)
Description: Percentage of patients with a complete response (CR) or partial response (PR) as assessed by Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1 (v1.1)
Time Frame: Approximately 3 years
Population: The clinical trial was terminated before participants were enrolled in Phase 2
Groups:
- Nanatinostat in Combination With Valganciclovir: Nanatinostat at the confirmed RP2D Valganciclovir at the confirmed RP2D
- Nanatinostat in Combination With Valganciclovir and Pembrolizumab: Nanatinostat at the confirmed RP2D Valganciclovir at the confirmed RP2D Pembrolizumab 200 mg IV every 3 weeks
Arm/Group | Nanatinostat in Combination With Valganciclovir | Nanatinostat in Combination With Valganciclovir and Pembrolizumab
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Incidence of Adverse Events
Description: Percentage of patients experiencing at least one treatment-emergent adverse event (AE), defined as those AEs with onset after the first dose of study drug or existing events that worsened after the first dose during the study
Time Frame: Approximately 3 years
Population: Safety analysis population, defined as all patients who received at least one dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Cohort 1 | Dose Cohort 2 | Dose Cohort 3 | Dose Cohort 4 | Dose Cohort 5 | Dose Cohort 6 | Dose Cohort 7
Number analyzed (Participants) | 3 | 4 | 3 | 3 | 4 | 3 | 6
Participants | 3 | 4 | 3 | 3 | 4 | 3 | 6

4. Secondary Outcome: Phase 2: Duration of Response (DOR)
Description: Interval of time from the date of first observed CR or PR to the date of documented disease progression or death due to any cause, whichever occurs first
Time Frame: Approximately 3 years
Population: The clinical trial was terminated before participants were enrolled in Phase 2
Arm/Group | Nanatinostat in Combination With Valganciclovir | Nanatinostat in Combination With Valganciclovir and Pembrolizumab
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Phase 2: Disease Control Rate (DCR)
Description: Percentage of patients having a CR, PR, or stable disease at any time during treatment
Time Frame: Approximately 3 years
Population: The clinical trial was terminated before participants were enrolled in Phase 2
Arm/Group | Nanatinostat in Combination With Valganciclovir | Nanatinostat in Combination With Valganciclovir and Pembrolizumab
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Phase 2: Progression-Free Survival (PFS)
Description: Interval of time from the start of study drug treatment to the date of first documented disease progression or death from any cause, whichever occurs first
Time Frame: Approximately 3 years
Population: The clinical trial was terminated before participants were enrolled in Phase 2
Arm/Group | Nanatinostat in Combination With Valganciclovir | Nanatinostat in Combination With Valganciclovir and Pembrolizumab
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Phase 2: Overall Survival (OS)
Description: Interval of time from the start of study drug treatment to date of death for any reason
Time Frame: Approximately 3 years
Population: The clinical trial was terminated before participants were enrolled in Phase 2
Arm/Group | Nanatinostat in Combination With Valganciclovir | Nanatinostat in Combination With Valganciclovir and Pembrolizumab
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Pharmacokinetic Parameter (Nanatinostat) - Time to Maximum Plasma Concentration [Tmax]
Description: Defined as the time required to reach peak plasma concentration [Cmax] after nanatinostat administration on Cycle 2 Day 1
Time Frame: Approximately 28 days following enrollment
Population: PK analysis population, defined as all patients who received at least 1 dose of nanatinostat on Cycle 2 Day 1 and had at least 1 valid PK concentration. The clinical trial was terminated before the outcome measure data were collected for Dose Cohort 6 and Dose Cohort 7.
Measure: Median (Full Range); unit: hours
Arm/Group | Dose Cohort 1 | Dose Cohort 2 | Dose Cohort 3 | Dose Cohort 4 | Dose Cohort 5 | Dose Cohort 6 | Dose Cohort 7
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 0 | 0
hours | 2 [1 to 4] | 1 [1 to 1] | 1 [1 to 2] | 4 [1 to 6] | 7 [2 to 8] |  |

9. Secondary Outcome: Pharmacokinetic Parameter (Ganciclovir) - Time to Maximum Plasma Concentration [Tmax]
Description: Defined as the time required to reach peak plasma concentration [Cmax] after valganciclovir administration on Cycle 2 Day 1
Time Frame: Approximately 28 days following enrollment
Population: PK analysis population, defined as all patients who received at least 1 dose of valganciclovir on Cycle 2 Day 1 and had at least 1 valid PK concentration. The clinical trial was terminated before the outcome measure data were collected for Dose Cohort 6 and Dose Cohort 7.
Measure: Median (Full Range); unit: hours
Arm/Group | Dose Cohort 1 | Dose Cohort 2 | Dose Cohort 3 | Dose Cohort 4 | Dose Cohort 5 | Dose Cohort 6 | Dose Cohort 7
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 0 | 0
hours | 2 [2 to 6] | 2 [2 to 2] | 2 [2 to 4] | 2 [2 to 4] | 2 [1 to 4] |  |

10. Secondary Outcome: Pharmacokinetic Parameter (Nanatinostat) - Maximum Plasma Concentration [Cmax]
Description: Defined as the peak plasma concentration [Cmax] after nanatinostat administration on Cycle 2 Day 1
Time Frame: Approximately 28 days following enrollment
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dose Cohort 1 | Dose Cohort 2 | Dose Cohort 3 | Dose Cohort 4 | Dose Cohort 5 | Dose Cohort 6 | Dose Cohort 7
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 0 | 0
ng/mL | 136 (137) | 391 (26.7) | 214 (44.8) | 96.1 (33.2) | 110 (53.8) |  |

11. Secondary Outcome: Pharmacokinetic Parameter (Ganciclovir) - Maximum Plasma Concentration [Cmax]
Description: Defined as the peak plasma concentration [Cmax] after valganciclovir administration on Cycle 2 Day 1
Time Frame: Approximately 28 days following enrollment
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dose Cohort 1 | Dose Cohort 2 | Dose Cohort 3 | Dose Cohort 4 | Dose Cohort 5 | Dose Cohort 6 | Dose Cohort 7
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 0 | 0
ng/mL | 4420 (3.49) | 5860 (32.1) | 5210 (80.9) | 7580 (32.6) | 4860 (27.2) |  |

12. Secondary Outcome: Pharmacokinetic Parameter (Nanatinostat) - Area Under the Plasma Concentration-Time Curve [AUC0-t]
Description: Defined as the area under the concentration-time curve from time 0 to the last measurable nanatinostat concentration on Cycle 2 Day 1
Time Frame: Approximately 28 days following enrollment
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Dose Cohort 1 | Dose Cohort 2 | Dose Cohort 3 | Dose Cohort 4 | Dose Cohort 5 | Dose Cohort 6 | Dose Cohort 7
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 0 | 0
ng*h/mL | 362 (82.2) | 751 (12.7) | 896 (39.0) | 416 (12.3) | 465 (67.2) |  |

13. Secondary Outcome: Pharmacokinetic Parameter (Ganciclovir) - Area Under the Plasma Concentration-Time Curve [AUC0-t]
Description: Defined as the area under the concentration-time curve from time 0 to the last measurable ganciclovir concentration on Cycle 2 Day 1
Time Frame: Approximately 28 days following enrollment
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Dose Cohort 1 | Dose Cohort 2 | Dose Cohort 3 | Dose Cohort 4 | Dose Cohort 5 | Dose Cohort 6 | Dose Cohort 7
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 0 | 0
ng*h/mL | 37200 (36.9) | 46700 (12.1) | 30900 (106) | 44400 (24.8) | 38200 (13.6) |  |

14. Secondary Outcome: Pharmacokinetic Parameter (Nanatinostat) - Half-Life of Nanatinostat [t1/2]
Description: Defined as the time required to reduce nanatinostat plasma concentration by 50% after nanatinostat administration on Cycle 2 Day 1
Time Frame: Approximately 28 days following enrollment
Population: PK analysis population, defined as all patients who received at least 1 dose of nanatinostat on Cycle 2 Day 1 and had at least 2 valid PK concentrations in the terminal elimination phase. The clinical trial was terminated before the outcome measure data were collected for Dose Cohort 6 and Dose Cohort 7.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Dose Cohort 1 | Dose Cohort 2 | Dose Cohort 3 | Dose Cohort 4 | Dose Cohort 5 | Dose Cohort 6 | Dose Cohort 7
Number analyzed (Participants) | 2 | 3 | 3 | 1 | 1 | 0 | 0
hours | 2.11 (0.136) | 1.43 (0.149) | 2.64 (1.90) | 2.76 (0) | 5.29 (0) |  |

15. Secondary Outcome: Pharmacokinetic Parameter (Ganciclovir) - Half-Life of Ganciclovir [t1/2]
Description: Defined as the time required to reduce ganciclovir plasma concentration by 50% after valganciclovir administration on Cycle 2 Day 1
Time Frame: Approximately 28 days following enrollment
Population: PK analysis population, defined as all patients who received at least 1 dose of valganciclovir on Cycle 2 Day 1 and had at least 2 valid PK concentrations in the terminal elimination phase. The clinical trial was terminated before the outcome measure data were collected for Dose Cohort 6 and Dose Cohort 7.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Dose Cohort 1 | Dose Cohort 2 | Dose Cohort 3 | Dose Cohort 4 | Dose Cohort 5 | Dose Cohort 6 | Dose Cohort 7
Number analyzed (Participants) | 2 | 3 | 2 | 3 | 4 | 0 | 0
hours | 6.88 (0.115) | 7.18 (1.48) | 5.64 (2.08) | 5.74 (0.601) | 6.07 (1.55) |  |

ADVERSE EVENTS:
Time Frame: Approximately 3 years
Arm/Group | Dose Cohort 1 | Dose Cohort 2 | Dose Cohort 3 | Dose Cohort 4 | Dose Cohort 5 | Dose Cohort 6 | Dose Cohort 7
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4 | 1/3 | 0/3 | 0/4 | 0/3 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/4 | 2/3 | 0/3 | 2/4 | 3/3 | 6/6
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 3/3 | 3/3 | 4/4 | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Cohort 1 (N=3) | Dose Cohort 2 (N=4) | Dose Cohort 3 (N=3) | Dose Cohort 4 (N=3) | Dose Cohort 5 (N=4) | Dose Cohort 6 (N=3) | Dose Cohort 7 (N=6)
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 2
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Creatinine renal clearance decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Electrocardiogram T wave abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Pneumonia aspiration (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Cohort 1 (N=3) | Dose Cohort 2 (N=4) | Dose Cohort 3 (N=3) | Dose Cohort 4 (N=3) | Dose Cohort 5 (N=4) | Dose Cohort 6 (N=3) | Dose Cohort 7 (N=6)
Blood creatinine increased (Investigations) | 1 | 2 | 0 | 1 | 3 | 3 | 6
Fatigue (General disorders) | 1 | 2 | 1 | 1 | 2 | 3 | 6
Nausea (Gastrointestinal disorders) | 1 | 2 | 2 | 1 | 1 | 3 | 5
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 1 | 1 | 1 | 3 | 5
Platelet count decreased (Investigations) | 1 | 1 | 0 | 1 | 2 | 3 | 6
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0 | 2 | 3 | 1 | 3
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0 | 2 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 1 | 2 | 2
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 3 | 0 | 2 | 1
White blood cell decreased (Investigations) | 0 | 1 | 0 | 2 | 0 | 2 | 2
Constipation (Gastrointestinal disorders) | 2 | 2 | 0 | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 3
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 2 | 1 | 0 | 3
Weight decreased (Investigations) | 0 | 0 | 0 | 1 | 3 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 2 | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 1 | 1
Creatinine renal clearance decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 2
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 2
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Contusion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Regurgitation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1

LIMITATIONS AND CAVEATS:
The study was prematurely terminated after the end of Phase 1b and did not proceed to Phase 2.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-09-22): https://cdn.clinicaltrials.gov/large-docs/77/NCT05166577/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-22): https://cdn.clinicaltrials.gov/large-docs/77/NCT05166577/SAP_001.pdf